CLINICAL TRIAL: NCT03279536
Title: Lactoferrin Versus Total Dose Infusion (TDI) For Treating Iron Deficiency Anemia in Pregnancy: Role of Nursing
Acronym: TDI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Howieda Fouly, PhD of Obstetric & Gynecologic Nursing, Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WHH
Record Dates: First submitted 2017-08-30; First posted 2017-09-12 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Lactoferrin

STUDY DESIGN:
Intervention Model Description: Group A will receive oral lactoferrin & group B will receive Total dose infusion
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Lactoferrin (Experimental): Group A is 120 mg of Oral lactoferrin for 4 weeks Intervention: The participants 66 will receive oral Lactoferrin 120mg for 4 weeks
  Interventions: Combination Product: Oral lactoferrin
- Total dose infusion (TDI) iron dextran (Active Comparator): Group B is a parenteral total dose infusion (TDI) of LMW iron dextran 20mg/kg body weight for 4 weeks Intervention: The participants 33 will receive parental iron 20mg/kg body weight for 4 weeks
  Interventions: Combination Product: TDI of LMW iron dextran

INTERVENTIONS:
Combination Product: Oral lactoferrin — Oral lactoferrin 120 mg twice /day and it's based on fast dissolving through direct swallowing per oral route with fruits flavor taste.
  Other Names: Oral Fizzing Lactoferrin
  Arms: Oral Lactoferrin
Combination Product: TDI of LMW iron dextran — Total Dose Infusion of LMW iron dextran up to 20mg/kg body weight is infused intravenously
  Other Names: Parental dextran
  Arms: Total dose infusion (TDI) iron dextran

SUMMARY:
This study consisted of 60 cases. All the cases of pregnant women are 4 months to 8 months of pregnancy. The cases divided into 30 pregnant women's were given iron supplementation without health education and another 30 were given iron supplementation and health education for comparison between them. Comparative between hemoglobin levels before and after medication. Treatment of iron deficiency anemia with iron supplementation received for one month.

DETAILED DESCRIPTION:
The investigator will divide the participants into two groups e.g. group (A) and group (B) according to Hemoglobin level and receiving of oral supplementation for IDA accompanied with health education in case of group (A) and without health education in case of group (B). Then the investigator asked patient to sign the document of her investigations result to receive iron supplementation.

* After that, the investigator observes hemoglobin's Level, when it less than >11g/dl, the patient will be the group (A) who will receive oral iron supplementation and health education.
* Group (B) who will receive Total Dose Infusion (TDI) without health education.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant Women aged >18 years
2. Hemoglobin<10g/dl
3. Gestational age between 14-28 weeks
4. Singleton pregnancy
5. Willingness to participate and signing the informed consent form

Exclusion Criteria:

1. Anemia predominantly caused by factors other than IDA (e.g. anemia with untreated B12 or foliate deficiency, hemolytic anemia),
2. Iron overload or disturbances in utilization of iron (e.g. hemochromatosis and haemosidrosis).
3. Decompensated liver cirrhosis and active hepatitis (ALAT>3 times upper limit of normal).
4. Active acute or chronic infections (assessed by clinical judgment supplied with white Blood Cells (WBC) and C - reactive protein (CRP).
5. Rheumatoid arthritis with symptoms or signs of active inflammation.
6. Multiple allergies.
7. Known hypersensitivity to parental iron or any recipients in the investigational drug products.
8. Erythropoietin treatment within 8 weeks prior to the screening visit.
9. Other iron treatment within 8 weeks prior to the screening visit.
10. Planned elective surgery during the study.
11. Participation in any other clinical within 3 months prior to the screening.
12. Any other medical condition e.g. malignancy, uncontrolled hypertension, unstable ischemic heart disease, or uncontrolled diabetes mellitus.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant female
Enrollment: 99 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
the change in Hb concentration | 4- 8 weeks
  measure the change in Hb concentration from baseline to week 4 after oral Lactoferrin treatment and relieve of symptoms of anemia

SECONDARY OUTCOMES:
measure the change in serum iron, serum ferritin | 4-8 weeks
  measure the change in serum iron, serum ferritin based on comparison between oral lactoferrin with health education & TDI from hospital routine care.

CONTACTS AND LOCATIONS:
Overall Officials: Warda Helmy, BSN, Principal Investigator — WHH
Locations (1):
- Women Health Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Publishing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3-6 months
Access Criteria: Introduction, Methodology, data analysis, Findings, Discussion & Conclusion